CLINICAL TRIAL: NCT05988944
Title: Which One is The Most Effective On The Hand Functions In Cerebral Palsy: Constraint-Induced Movement Therapy or Constraint-Induced Movement Therapy With Virtual Reality? A Randomized Controlled Trial.
Brief Title: The Hand Functions In Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Cetin Sayaca, Principal Investigator; Assos. Prof., Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIMT vs VR
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy; Hand Functions
Keywords: Hand Functions; Virtual Reality; Constraint-Induced Movement Therapy; Cerebral Palsy; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional techniques (Active Comparator): TT was planned according to the child's hand that was needed. Neurodevelopmental facilitation techniques (Bobath therapy), stretching, and grasping types (cylindrical, spherical, hook, key, fingertip, lateral) were used in hands therapy for 45 minutes two days in a week for all children who were accepted to participate in this study.
  Interventions: Other: TT
- traditional therapy with constraint induced movement therapy (Experimental): The sling was put on the child's non-paretic arm to apply CIMT. The around of the sling was sewn except the elbow and secured snugly to the trunk with a waist strap to prevent assisting the affected hand during the application of CIMT. However, children with CP who were in the this group used the sling for three hours in daily activity, playing, etc. at home. The CIMT was given as a home program and monitorization was done by the follow-up form every week with no therapy during the weekend.
  Interventions: Other: TT+CIMT
- traditional therapy with constraint induced movement therapy and virtual reality (Experimental): After the TT session, a child with CP used the sling for 45 minutes at the rehabilitation center with VR therapy. VR therapy with CIMT was used in hands therapy for 45 minutes at two days a week after TT. During the VR therapy, the child was encouraged verbally to play X-box.The X-box Kinect 360 (by the Microsoft corporation) was used for VR therapy. It has a kinetic sensor that perceives the movement of the child with CP. The child's movement can be seen through the monitor in real time. VR does not need special buttons to play. Therefore, a child with CP who had impaired fine motor skills and dexterity can play easily.
  Interventions: Other: TT+CIMT+VR

INTERVENTIONS:
Other: TT+CIMT+VR — TT: Traditional Techniques CIMT: constraint-induced movement therapy VR: virtual reality
  Arms: traditional therapy with constraint induced movement therapy and virtual reality
Other: TT+CIMT — TT: Traditional Techniques CIMT: constraint-induced movement therapy
  Arms: traditional therapy with constraint induced movement therapy
Other: TT — TT: Traditional Techniques
  Arms: Traditional techniques

SUMMARY:
The hand motor functions are very important in the daily life activities, educational, and social participation of children. Losing The hand motor functions limit these activities and participation. Constraint-induced movement therapy (CIMT) or virtual reality (VR) therapy has often been preferred to improve the hand's motor functions.

DETAILED DESCRIPTION:
CIMT and VR are used to improve the motor functions of the hand in cerebral palsy (CP). The aim of this study was to compare the effects of CIMT-VR use and only CIMT use on hand functions in children with hemiparetic cerebral palsy. Hand function and performance were evaluated with the Jebsen-Taylor and Moberg pick-up tests. All evaluations were made twice; before the first therapy and after six weeks. Children with hemiparetic CP were divided into three groups randomly (Traditional techniques (TT), TT+CIMT, and TT+CIMT+VR).

ELIGIBILITY:
The inclusion criteria of the study were determined to be

* aged 8 to 18 years,
* diagnosed with hemiparetic CP,
* being level 2 or 3 according to the gross motor function measurement scale and the manual ability classification system.

The exclusion criteria of the study were,

* severe cognitive dysfunction that rendered them unable to perform simple tasks (e.g., reaching, grasping),
* having pharmacologic medicine for spasticity,
* having botulinum toxin A injections in the last 6 months,
* having upper extremity surgery,
* having visual and/or auditory problems which affect therapy or evaluation.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
The Jebsen-Taylor Test | this evaluation was done twice; before the first therapy and after six weeks by the same physiotherapist.
  The Jebsen-Taylor Test is a reliable tool that evaluates the hand function of children with CP. The test includes seven items. These items are; writing a 24-letter sentence, turning over five cards, picking up small objects (two pieces of pennies/bottle caps/paperclips), simulated feeding (using a teaspoon and five kidney beans), stacking four checkers, picking up and moving five large empty tin boxes and then five large full boxes. During the assessment, the child with CP was seated in front of a table and test was performed by hemiparetic hand. Time was recorded on each item by stopwatch. The total score was calculated by collecting all items' time.
Moberg pick-up test | this evaluation was done twice; before the first therapy and after six weeks by the same physiotherapist.
  To evaluate the functional performance of the hemiparetic hand Moberg pick-up test (MPUT) was used. MPUT consists of twelve items which are a wing nut, screw, key, nail, ₺1 coin, 50 kurus coin, washer, safety pin, paper clip, large and medium-sized hexagonal nut, and small square nut. The plastic container (60x30 cm) was placed lengthwise about 15 cm from the edge of the table on the opposite side of the items. The child was seated in a chair. The hemiparetic hand of children with CP was put on the same side as the 12 items which were randomly placed on the table. Children with CP were ordered to pick up the items one at a time and place them into the plastic container as fast as possible. The time was recorded with a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Esin KADIKOYLU, Pt, Study Chair — Uskudar University; Eren DEMIRAYAK, Pt, Study Chair — Uskudar University; Cetin Sayaca, Assoc. Prof., Principal Investigator — Uludag University
Locations (1):
- Uskudar Universty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliott C, Reid S, Hamer P, Alderson J, Elliott B. Lycra((R)) arm splints improve movement fluency in children with cerebral palsy. Gait Posture. 2011 Feb;33(2):214-9. doi: 10.1016/j.gaitpost.2010.11.008. Epub 2010 Dec 4. PMID 21131201
- [Background] Hoare BJ, Wallen MA, Thorley MN, Jackman ML, Carey LM, Imms C. Constraint-induced movement therapy in children with unilateral cerebral palsy. Cochrane Database Syst Rev. 2019 Apr 1;4(4):CD004149. doi: 10.1002/14651858.CD004149.pub3. PMID 30932166
- [Background] Sakzewski L, Ziviani J, Boyd R. Systematic review and meta-analysis of therapeutic management of upper-limb dysfunction in children with congenital hemiplegia. Pediatrics. 2009 Jun;123(6):e1111-22. doi: 10.1542/peds.2008-3335. Epub 2009 May 18. PMID 19451190
- [Background] Brady K, Garcia T. Constraint-induced movement therapy (CIMT): pediatric applications. Dev Disabil Res Rev. 2009;15(2):102-11. doi: 10.1002/ddrr.59. PMID 19489088
- [Background] Jung SH, Song SH, Kim SD, Lee K, Lee GC. Does virtual reality training using the Xbox Kinect have a positive effect on physical functioning in children with spastic cerebral palsy? A case series. J Pediatr Rehabil Med. 2018;11(2):95-101. doi: 10.3233/PRM-160415. PMID 30010148